CLINICAL TRIAL: NCT05420948
Title: A Phase II Study of Pembrolizumab in Combination With Circulating Tumor DNA Response-Adaptive Pulsed Chemotherapy in Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma: The SINERGY Trial (Squamous Cell Carcinoma of Head and Neck Response-Guided Therapy)
Brief Title: A Study of Pembrolizumab in Combination With Chemotherapy for Head and Neck Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB22-0288
Record Dates: First submitted 2022-06-13; First posted 2022-06-15 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Head and Neck Neoplasms; Head Cancer; Throat Carcinoma
Keywords: head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Participants Who Receive Pembrolizumab (Alone) (Experimental): Participants in this group will receive pembrolizumab 200 mg through an intravenous (IV) needle inserted into the arm. Medications will be given on day 1 of each 21-day cycle for two cycles..
  Interventions: Drug: Pembrolizumab
- Group 2: Participants Who Receive Pembrolizumab + Chemotherapy with Carboplatin and Paclitaxel (Experimental): Participants in this group will receive 200 mg of pembrolizumab through an intravenous (IV) needle inserted into the arm plus chemotherapy with carboplatin (AUC 6) on day 1 and paclitaxel (200 mg) on day 1 of each 21-day cycle for two cycles.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab — A drug that binds to a protein called programmed cell death 1 (PD-1) to help immune cells kill cancer cells better. Pembrolizumab is used to treat many different types of cancer.
  Other Names: KEYTRUDA
Drug: Carboplatin — A chemotherapy drug used to treat cancer.
  Other Names: Paraplatin
  Arms: Group 2: Participants Who Receive Pembrolizumab + Chemotherapy with Carboplatin and Paclitaxel
Drug: Paclitaxel — A chemotherapy drug used to treat cancer.
  Other Names: Taxol
  Arms: Group 2: Participants Who Receive Pembrolizumab + Chemotherapy with Carboplatin and Paclitaxel

SUMMARY:
By doing this study, the research team would like to learn if using a blood test that measures the amount of tumor DNA in blood can help guide how to use chemotherapy combined with immunotherapy for individuals with head and neck cancer. Using this blood test, the research team hopes to learn if intermittent (occasional) chemotherapy added to immunotherapy will work better than immunotherapy alone. Participation in this research will last about two years.

DETAILED DESCRIPTION:
By doing this study, the research team hopes to learn if using a blood test that measures the amount of tumor DNA in blood can help guide how to use chemotherapy combined with immunotherapy for individuals with head and neck cancer. Using this blood test, the research team hopes to learn if intermittent (occasional) chemotherapy added to immunotherapy will work better than immunotherapy alone. Participation in this research will last about two years.

The purpose of this research is to gather information on how well immunotherapy with intermittent chemotherapy guided by measurements of tumor DNA in blood will work and to learn about the safety and effectiveness of this new treatment strategy. All of the drugs used in this trial are approved by the US Food and Drug Administration (FDA); however, they are being combined in a new way based on changes in tumor DNA in the participant's blood which can only be done in a research study.

ELIGIBILITY:
Inclusion Criteria:

* Have clinically confirmed head and neck cancer that is recurrent (comes back/returns to the body) or metastatic (spreads to other parts of the body).
* Participants should not have had prior systemic therapy administered in the recurrent or metastatic setting. Systemic therapy which was completed more than 3 months prior to signing consent if given as part of multimodal treatment for locally advanced disease is allowed.
* Greater than or equal to 18 years old.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Have measurable disease based on RECIST 1.1 as determined by the site. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Participants must have normal organ and marrow function as defined by clinical lab values.
* Participants must have provided tissue for programmed cell death ligand 1 (PD-L1) biomarker analysis from a core or excisional biopsy (fine needle aspirate is not adequate). Repeat samples may be required if adequate tissue is not provided. A newly obtained biopsy (within 90 days prior to start of study treatment) is strongly preferred, but an archival sample is acceptable.
* Measurable disease (either primary site and/or nodal disease) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
* Participants must sign a study-specific informed consent form prior to study entry. Participants should have the ability to understand and the willingness to sign a written informed consent document.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
* Women must not be breastfeeding.
* Women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment.
* Men who are sexually active with women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s).

Exclusion Criteria:

* Has disease that is suitable for local therapy administered with curative intent.
* Has progressive disease (PD) within three (3) months of completion of curatively intended systemic treatment for locoregionally advanced head and neck cancer.
* Participants who are receiving any other investigational agents.
* Participants in whom signatera ctDNA is not measurable at baseline.
* Has had radiation therapy (or other non-systemic therapy) within 2 weeks prior to enrollment or patient has not fully recovered (i.e., ≤Grade 1 or at baseline) from adverse events due to a previously administered treatment.

  * Note: Participants with ≤Grade 2 neuropathy, ≤Grade 2 alopecia, are an exception to this criterion and may qualify for the study.
  * Note: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Active, known, or suspected, autoimmune or inflammatory disorders requiring immunosuppressive therapy, with the exception of low-dose prednisone (<= 10mg or equivalent). The following are exceptions to these criteria:
* Participants with vitiligo or alopecia.
* Participants with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.
* Any chronic skin condition that does not require systemic treatment.
* Has a life expectancy of less than 3 months and/or has rapidly progressing disease (e.g. tumor bleeding, uncontrolled tumor pain) in the opinion of the treating investigator.
* Participants with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥ 3 years.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Has had an allogeneic tissue/solid organ transplant.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab or other agents used in study.
* Has received prior therapy with an anti-PD1(anti-programmed cell death protein1) therapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Pregnant women are excluded from this study because pembrolizumab is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab, breastfeeding should be discontinued if the mother is treated with pembrolizumab. These potential risks may also apply to other agents used in this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with pembrolizumab, carboplatin, and paclitaxel. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Has known active Hepatitis B or Hepatitis C. However, if eradicated participant is eligible.
* Has a history of active infection requiring systemic therapy.
* Has received a live vaccine within 28 days of planned start of study therapy. Note: Vaccines for COVID-19 are allowed except for any live vaccine that may be developed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate of Participants as Assessed by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). | 2 years
  Overall response rate with pembrolizumab in combination with circulating tumor DNA (ctDNA) chemotherapy among subjects with head and neck cancer. Response rate will be defined as the proportion of participants with a complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
The Rate of Adverse Events Reported Among Study Participants Receiving Pembrolizumab + Chemotherapy Compared to The Rate of Adverse Events Reported Among Participants Who Received Pembrolizumab + Chemotherapy in a Related Study | 2 years
  The rate of adverse events (Grade 3 of higher) reported among participants who receive pembrolizumab + chemotherapy compared to the rate of adverse events (Grade 3 or higher) reported among participants who received pembrolizumab +chemotherapy in a previous related study called Keynote-48. Adverse events will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.
Progression Free Survival of Participants Receiving Pembrolizumab + Chemotherapy | 2 years
  Progression Free Survival of pembrolizumab combination with circulating tumor DNA (ctDNA) response-adaptive pulsed chemotherapy among participants. Progression free survival will be defined as the time from date of first dose of study drug to date of documented progressive disease (PD) based on Response Evaluation Criteria in Solid Tumors version 1.1 ( RECIST v1.1 )or death, whichever occurs first.
Overall Survival of Participants Receiving Pembrolizumab + Chemotherapy | 2 years
  The overall survival of pembrolizumab in combination with circulating tumor DNA (ctDNA) response-adaptive pulsed chemotherapy in participants with head and neck cancer. Overall survival will be defined as the time from the date of first dose of study drug to the date of death.
Duration of Response of Participants Receiving Pembrolizumab + Chemotherapy | 2 years
  The duration of response (DoR) of pembrolizumab in combination with circulating tumor DNA (ctDNA) response-adaptive pulsed chemotherapy in participants with head and neck cancer. Duration of response will be defined as the time from date of first documented response to the date of documented progressive disease or death, based on Response Evaluation Criteria in Solid Tumors version 1.1 ( RECIST v1.1).
The Rate of Adverse Events Reported Among Study Participants Receiving Pembrolizumab + Chemotherapy | 2 years
  The rate of adverse events reported among participants who receive pembrolizumab in combination with chemotherapy as assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.
Rate of Adverse Events Leading to Discontinuation or Death Among Participants | 2 years
  Rate of adverse events leading to discontinuation or death among participants as assessed by Common Criteria Terminology for Adverse Events (CTCAE v. 5.0).
Proportion of Participants who Receive a Lower Dose of Study Drugs After Treatment with Pembrolizumab + Chemotherapy | 2 years
  Proportion of participants who begin to receive a lower dose of study drugs (known as a "de-escalated" dose) based on decreases in circulating tumor DNA (ctDNA) from pembrolizumab and chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Rosenberg, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States